CLINICAL TRIAL: NCT05586256
Title: Ultra-hypofractionated Adjuvant Radiotherapy After Breast Conserving Surgery in Breast Cancer Patients
Brief Title: Ultra-hypofractionated Radiotherapy in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Cynthia Aristei, Professor, University Of Perugia
Other Study IDs: FAST-F-PG01
Record Dates: First submitted 2022-10-05; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Female Breast Cancer
Keywords: early stage breast cancer; breast conserving surgery; ultra-hypofractionated whole breast irradiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: ultra-hypofractionated whole breast irradiation — All enrolled patients will be treated with an ultra-ipofractionated whole breast irradiation schedule (26 Gy delivered in 5 consecutive fractions, single dose 5.2 Gy), according to FAST-Forward trial. Whole bresat irradiation should be followed or not by a tumor bed boost (sequential: 7.6 Gy in 2 consecutive fractions, single dose 3.8 Gy or simultaneous intergrated boost: 30 Gy in 5 consecutive fractions, single dose 6 Gy). Either three-dimensional conformal radiotherapy (3DCRT), intensity-modulated radiotherapy (IMRT), volumetric modulated arc therapy (VMAT) or helicoildal techniques are allowed. Breath control techniques may be used at the discretion of each partecipating centre.
  Main exclusion critereria are mastectomy and regional nodal irradiation. Neoadjuvant and/or adjuvant systemic therapies are allowed.

SUMMARY:
The present multicenter, retrospective and prospective observational study, aims to evaluate an ultra-hypofractionated whole breast irradiation schedule (WBI, 26 Gy in 5 fractions), in order to confirm literature data (FAST-F study) in the clinical practice.

Patient population included women affected by early stage breast cancer (BC), both invasive and ductal carcinoma in situ, receiving ultra-hypofractionated WBI (with or without a tumor bed boost) after breast conserving surgery (BCS). Main exclusion criteria are mastectomy and regional nodal irradiation. Neoadjuvant and/or adjuvant systemic therapies are allowed. The primary otcome is acute and chronic toxicity evaluation. Secondary outcomes are: overall servival (OS), disease-free survival (DFS), rates of local and loco-regional recurrences, distant metastasis occurrence, cosmetic outcome and quality of life (QoL) assessment. Acute and late toxicities will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0. Cosmetic assessment will be graded according to the Harvard scale. Frontal photographs of both breasts will be used to evaluate toxicity and cosmetic results. For QoL assessment the EORTC (European Organisation for Research and Treatment of Cancer), QLQ-C30 and EORTC-QLQ-BR23 questionnaires will be administered.

DETAILED DESCRIPTION:
The present multicenter retrospective and prospective observational study aims to evaluate feasibility, toxicity, efficacy, cosmetic outcome and QoL in early stage BC patients treated with BC followed by ultra-hypofractionated WBI (with or without a tumor bed boost). This study was designed to confirm literature data (FAST-Forward trial) in the clinical practice ("real life"study). All enrolled patients will be treated with an ultra-hypofractionated WBI schedule (26 Gy delivered in 5 consecutive fractions, single dose 5.2 Gy), according to FAST-Forward trial. Whole breast irradiation should be followed or not by a tumor bed boost (sequential: 7.6 Gy in 2 consecutive fractions, single dose 3.8 Gy or simultaneous intergrated boost: 30 Gy in 5 consecutive fractions, single dose 6 Gy). Either three-dimensional conformal radiotherapy (3DCRT), intensity-modulated radiotherapy (IMRT), volumetric modulated arc therapy (VMAT) or helicoildal techniques are allowed. Breath control techniques may be used at the discretion of each partecipating centre. Main exclusion criteria are mastectomy and needs for regional nodal irradiation. Neoadjuvant and/or adjuvant systemic therapies are allowed.

The primary outcome of this study is acute and chronic toxicity evaluation. Secondary outcomes are: OS, DFS, rates of local and loco-regional recurrence, distant metastasis occurence, cosmetic outcome and QoL assessment. Acute and late toxicities will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0 at each follow-up visit.

Regarding prospectively enrolled patient cosmetic assessment will be graded (by the physician and the patient) according to the Harvard scale and performed before the start of radiotherapy (RT), 6 months and 1, 2 and 5 years after the end of RT; frontal photographs of both breasts will be taken before the start of R, 6 months and 1, 2 and 5 years after the end of RT. In particular, two photographs will be taken of the patient's trunk region, one with the hands resting on the hips, the other with the arms raised above the head (avoiding patients face). Photographic documentation will be evaluated according to the consensus scoring method described by Haviland et al. For QoL assessment the EORTC (European Organisation for Research and Treatment of Cancer), QLQ-C30 and EORTC-QLQ-BR23 will be administered before the start of RT,1 month after the end of RT and then at 1, 2 and 5 years after the end of RT.

Follow-up visits are scheduled as follows: one month after the end of RT and then every 4-6 months for 5 years. Laboratory test (blood count, biochemical, with or without CEA and Ca15.3), mammography and breast ultrasound scans will be scheduled 4-6 months after the end of RT and then yearly. Additional exams will be prescribed during the follow up in order to detected any disease reccurence.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age ≥ 18 years.
* Early stage breast cancer treated with breast conserving surgery
* Whole breast irradiation without regional nodal irradiation
* Infiltrating carcinomas
* CDIS
* Written informed consent

Exclusion Criteria:

* Age<18 years.
* Regional nodal radiotherapy.
* Distant metastases.
* Previous history of malignancy except basaloid skin tumours and CIN. Previous history of breast cancer is not an exclusion criteria if treated with curative intent and if patient is disease free at least 5 years from diagnosis.
* Presence of absolute radiotherapy contraindications (pregnancy, inability to maintain the correct treatment position) and relative radiotherapy contraindications (connective tissue diseases including rheumatoid arthritis, scleroderma, systemic lupus erythematosus, dermatomyositis and vasculitis, especially if the disease is in an active phase)
* Patient's refusal to use data for research purposes.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by early stage breast cancer (both invasive and ductal carcinoma in situ) receiving ultra-hypofractionated whole breast irradiation (with or without a tumor bed boost) after breast conserving surgery. Main exclusion critereria are mastectomy and regional nodal irradiation .Neoadjuvant and/or adjuvant systemic therapies are allowed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 1-6 months after RT
  Evaluation of acute toxicity to confirm the results obtained in the prospective randomized FAST-Forward study. Acute toxicity will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0
Late toxicity | from 6 months after RT to 60 months
  Evaluation of chronic late toxicity to confirm the results obtained in the prospective randomized FAST-Forward study. Late will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0

SECONDARY OUTCOMES:
overall survival | 1 month after RT and then every 4-6 months for 5 years
  overall survival
disease-free survival | 1 month after RT and then every 4-6 months for 5 years
  disease-free survival
rates of local and loco-regional recurrence | 1 month after RT and then every 4-6 months for 5 years
  rates of local and loco-regional recurrence
distant metastasis occurence | 1 month after RT and then every 4-6 months for 5 years
  distant metastasis occurence
cosmetic outcome | at baseline and then after 6 months and then 1, 2 and 5 years
  Breast cosmetic result will be graded according to Harvard scale of breast cosmesis (1. Excellent - 2. Good - 3. Fair - 4. Poor)
QoL assessment | at baseline and then after 6 months and then 1, 2 and 5 years
  EORTC QLQ-C30
QoL assessment | at baseline and then after 6 months and then 1, 2 and 5 years
  EORTC-QLQ-BR23
photographic assessment | at baseline and then after 6 months and then 1, 2 and 5 years
  consensus scoring method described by Haviland et al.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aristei, MD, Principal Investigator — Radiation Oncology Section, Department of Medicine and Surgery, University of Perugia
Locations (1):
- Radiation Oncology Section, Department of Medicine and Surgery, University of Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mariam NBG, Song YP, Joseph N, Hoskin P, Reeves K, Porta N, James N, Choudhury A. Hypofractionation: less is more? Oncotarget. 2021 Aug 17;12(17):1729-1733. doi: 10.18632/oncotarget.28023. eCollection 2021 Aug 17. PMID 34434502
- [Background] Haviland JS, Ashton A, Broad B, Gothard L, Owen JR, Tait D, Sydenham MA, Yarnold JR, Bliss JM. Evaluation of a method for grading late photographic change in breast appearance after radiotherapy for early breast cancer. Clin Oncol (R Coll Radiol). 2008 Sep;20(7):497-501. doi: 10.1016/j.clon.2008.03.017. Epub 2008 May 27. PMID 18502105
- [Background] Harris JR, Levene MB, Svensson G, Hellman S. Analysis of cosmetic results following primary radiation therapy for stages I and II carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1979 Feb;5(2):257-61. doi: 10.1016/0360-3016(79)90729-6. No abstract available. PMID 110740